CLINICAL TRIAL: NCT06961955
Title: FAST NOVEMBER: A Phase II Randomized Trial of a 5 vs. 9-day Course of Whole Breast Radiotherapy With Boost for Early-stage Breast Cancer
Brief Title: 5 vs. 9-day Course of Whole Breast Radiotherapy With Boost for Early-stage Breast Cancer
Acronym: FAST NOVEMBER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI189208
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Invasive Carcinoma of Breast; Ductal Breast Carcinoma in Situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Radiotherapy

STUDY DESIGN:
Masking Description: Study will have no masking as the treating investigator and patient will need to know their radiation schedule for accurate treatment planning.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 5 fractions of radiotherapy (Arm 1) (Experimental)
  Interventions: Radiation: Radiation Therapy
- 9 fractions of radio therapy (Arm 2) (Active Comparator)
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Undergo hypofractionated radiation therapy

SUMMARY:
The goal of this study is to evaluate 5 days vs. 9 days of whole breast radiation.

ELIGIBILITY:
Inclusion Criteria:

* Female participant aged ≥ 18 years.

  --Participants must have at least one of the following risk factors:
  * Grade 3 invasive histology
  * Estrogen receptor positivity less than 5%
  * Lymphovascular invasion
  * Invasive margins <2mm on surgical pathology
  * DCIS final positive margin
  * Extensive intraductal component
  * Age ≤ 50 years
  * Tumor size > 2 cm
* Histologically confirmed invasive carcinoma or Ductal Carcinoma In Situ (DCIS) of the breast.
* Breast cancer stage (AJCC v8) T0-3, N0, M0. T0 N0 is allowed if whole breast radiation is recommended by the treating physician.
* Lumpectomy within 84 days of the start of radiation.
* ECOG Performance Status ≤ 2, or KPS ≥ 50
* Negative inked histologic margins from lumpectomy, with the exception of a focus of positive margin at the pectoralis fascia.
* Negative pregnancy test for participants of childbearing potential, evidence of permanent surgical sterilization, or post-menopausal status. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * < 50 years of age:

    * Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and
    * Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution
  * ≥ 50 years of age:

    * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments; or
    * Had radiation-induced menopause with last menses >1 year ago; or
    * Had chemotherapy-induced menopause with last menses >1 year ago
* Sexually active participants of childbearing potential must agree to use highly effective method of contraception (defined in Section 5.4.1) during the course of radiation and for 30 days after radiation.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Bilateral breast cancer.
* Prior radiation therapy to the chest.
* Prior chemotherapy.
* Recurrent disease.
* Known metastases or node positive.
* Major chest surgery which is expected to impact study participation 8 weeks prior to starting study drug.
* Prior breast malignancy in either breast.
* The diagnosis of any other malignancy which, in the opinion of the Investigator, is likely to negatively impact the subject's safety or ability to participate in the study.
* Current evidence of uncontrolled, significant intercurrent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association Class III or IV, unstable angina pectoris, serious cardiac arrhythmias.
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic events, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 3 months before the first dose.
  * Any other condition that would, in the Investigator's judgment, contraindicate the participant's participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g., infection/inflammation, intestinal obstruction, unable to swallow, social/ psychological issues, etc.)
* Significant post lumpectomy complications requiring an unplanned re-operation for surgical complications or admission for IV antibiotics. Re-operation for margins evaluation or nodal evaluation is acceptable. Draining of a seroma is not considered a complication unless it has become infected.
* Breast neuroendocrine carcinoma or sarcoma histology.
* Radiation sensitizing disease or condition (e.g. connective tissue disease, li fremani, etc.).
* Medical, psychiatric, cognitive, or other conditions that may compromise the participant's ability to understand the participant information, give informed consent, comply with the study protocol or complete the study.
* Participants receiving concurrent radiation sensitizing medications or therapies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participant aged ≥ 18 years
Enrollment: 144 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2033-05 (Estimated)

PRIMARY OUTCOMES:
24-month Mean breast overall satisfaction Breast - Q scores with 5 fractions of radiation is non-inferior in patient reported outcomes. | 3 years
  To evaluate non-inferiority of 24-month Breast-Q satisfaction with breast score with 5 versus 9 fractions of radiation.

SECONDARY OUTCOMES:
Evaluate acute and late radiation-related adverse events (AEs) and serious adverse events (SAEs) between the two arms, characterized by type | 5 years
  To estimate the incidence of acute and late radiation complications between the two arms, based on CTCAE 5.0 toxicity.
Evaluate acute and late radiation-related adverse events (AEs) and serious adverse events (SAEs) between the two arms, characterized by severity (as defined by the NIH CTCAE, version 5.0) | 5 years
  To estimate the incidence of acute and late radiation complications between the two arms, based on CTCAE 5.0 toxicity.
Evaluate acute and late radiation-related adverse events (AEs) and serious adverse events (SAEs) between the two arms, characterized by seriousness | 5 years
  To estimate the incidence of acute and late radiation complications between the two arms, based on CTCAE 5.0 toxicity.
Evaluate acute and late radiation-related adverse events (AEs) and serious adverse events (SAEs) between the two arms, characterized by duration | 5 years
  To estimate the incidence of acute and late radiation complications between the two arms, based on CTCAE 5.0 toxicity.
Evaluate acute and late radiation-related adverse events (AEs) and serious adverse events (SAEs) between the two arms, characterized by relationship to study treatment. | 5 years
  To estimate the incidence of acute and late radiation complications between the two arms, based on CTCAE 5.0 toxicity.
Evaluate non-inferiority of local and local regional recurrence rate in the treatment arms. | 8 years
  To evaluate non-inferiority of the local and local regional recurrence rate between the two arms.
Evaluate non-inferiority of a change in cosmetic scores in the treatment arms with pre-radiation scores to post 24-month scores using the UK photographic assessment and EORTC scales. | 5 years
  To evaluate non-inferiority of the breast photographic cosmetic outcomes of the UK and EORTC scales
60-month mean breast overall satisfaction Breast-Q scores with 5 fractions of radiation is non-inferior in patient reported outcomes. | 5 years
  To evaluate non-inferiority of the mean Breast-Q scores with 5 fractions of radiation at 60 months.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R. Poppe, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No